CLINICAL TRIAL: NCT07158580
Title: Opti Gait Wearable Gait Tracker: Pilot Trial l With Healthy Older Adults
Brief Title: Opti Gait Wearable Gait Tracker
Status: Not yet recruiting | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2025-1220; R33AG061699-06 (NIH); ENGR/ELECTRICAL & COMPUTER ENG (Other: UW Madison); AS (Other: UW Madison); Protocol Version 8/13/2025 (Other: UW Madison)
Record Dates: First submitted 2025-08-28; First posted 2025-09-08 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-08

CONDITIONS: Seniors

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- No gait or mobility issues: Participants aged 65 or older who are able to walk for at least 10 minutes and can walk up and down a flight of stairs
  Interventions: Device: Gait Tracker

INTERVENTIONS:
Device: Gait Tracker — Opti Gait is a wearable gait tracker
  Other Names: OptiGait Wearable Gait Tracker

SUMMARY:
The purpose of this observational study is to test a shoe mounted gait monitoring device that was refined with the input of older adults and assess the efficacy of the refinements through a series of tests that involve walking with and without the device.

DETAILED DESCRIPTION:
In this testing, researchers seek to validate the precision, accuracy and robustness of the community-corefined device with healthy older adults, aged 65 years and above, by conducting walking tests on a state of the art GaitRite gaitmat to assess various gait metrics and on a flight of stairs to assess gait height. Following this, researchers will conduct a semi structured interview that will comprise a series of yes/no questions and open ended questions to understand the efficacy of the refinements and further refinement directions.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 years and older
* Able to speak and understand English,
* Able to provide consent

Exclusion Criteria:

* Current or recent (< 1 year) major psychiatric condition
* Significant medical condition such that usability evaluation could pose substantial health or safety risk
* Individuals with an activated power of attorney will be excluded from the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Adults aged 65 years and older that have low technology literacy, and are from underserved urban and rural areas.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Change in walking speed | 3 hours
  Participants will walk 4 meters with and without the shoe mounted device to assess the change in walking speed
Change in natural gait | 3 hours
  Participants will walk on a gait mat to assess natural gait, and then will walk on the gait mat wearing the device to assess the change in natural gait. Gait metrics captured by OptiGait will be compared with those captured by GaitRite to understand accuracy and precision.
Gait height | 3 hours
  Participants will climb a flight of five stairs, wearing the device, to measure gait height.

CONTACTS AND LOCATIONS:
Overall Officials: Jayer Fernandes, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin - Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes